CLINICAL TRIAL: NCT00235300
Title: An Open-Label Prospective, Randomized, Multicenter Phase II Comparative Trial of Thymoglobulin® Versus Simulect® for the Prevention of Delayed Graft Function and Acute Allograft Rejection in Renal Allograft Recipients
Brief Title: An Open-label, Prospective, Randomized, Multi-center, Phase II Comparative Trial of Thymoglobulin Versus Simulect for the Prevention of Delayed Graft Function and Acute Allograft Rejection in Renal Allograft Recipients.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SMC-101-1010
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Cadaveric Donor Renal Transplantation; Acute Renal Allograft Rejection; Induction Therapy
Keywords: Anti-T cells antibodies; Cadaveric Donor Renal Transplantation; Acute Renal Allograft Rejection; Induction Therapy
MeSH Terms: interventions — thymoglobulin; Antilymphocyte Serum; Basiliximab

ARMS (2):
- 1 Control (Active Comparator): Simulect (basiliximab)
  Interventions: Drug: Simulect (basliximab)
- 2 (Experimental): Thymoglobulin (anti-thymocyte globulin (rabbit))
  Interventions: Biological: Thymoglobulin [Anti-thymocyte Globulin (rabbit)]

INTERVENTIONS:
Biological: Thymoglobulin [Anti-thymocyte Globulin (rabbit)] — 1.5 mg/kg per day, for a maximum of 5 doses
  Arms: 2
Drug: Simulect (basliximab) — 20 mg per day on 2 days
  Arms: 1 Control

SUMMARY:
A multicenter clinical study comparing event-free survival at 6 months after transplant between Thymoglobulin-treated and Simulect-treated adult kidney transplant patients. Patients received Thymoglobulin or Simulect from Day 0 through Day 4. Day 0 was considered the day of the transplant procedure.

Subjects meeting all inclusion and exclusion criteria were eligible to participate in this study. The treatment assignment was random and not chosen by the subject or their physician.

Subjects were monitored during treatment with Thymoglobulin and during the transplant hospitalization. Additional subject monitoring occurred up to 12 months after transplant.

278 study subjects were enrolled at 28 transplant centers in the United States and Europe.

ELIGIBILITY:
Inclusion Criteria:

* Patient greater than or equal to 18 years old.
* Patient is classified as "high risk" for acute allograft rejection of DGF. Must have had at least 1 donor or 1 recipient variable for high risk.
* Patient will be a recipient of a solitary cadaveric renal allograft.
* Women of childbearing potential must have had a negative pregnancy test (serum or urine).
* Man or woman agrees to practice medically acceptable contraception (i.e. barrier or pharmacologic) for a minimum of 3 months following study drug administration. In addition, women were recommended to practice contraception for 1 year following transplantation, or per local standard.
* Patient agrees to participate in the study and sign an informed consent.
* Patient has no known contraindication to the administration of rabbit anti-thymocyte globulin or basiliximab. Patient has no history of hypersensitivity to basiliximab.
* Patient is dialysis-dependent at the time immediately prior to transplantation.

Exclusion Criteria:

* Patient has received an investigational medication within the past 30 days.
* Patient has a history of malignancy within 2 years, with the exception of adequately treated localized squamous basal cell carcinoma of the skin without evidence of recurrence.
* Patient is currently abusing drugs or alcohol.
* Patient is known or suspected to have an active infection or be seropositive for hepatitis B surface antigen (HBsAg), hepatitis C (HCV), or human immunodeficiency virus (HIV).
* Patient is a multiple organ transplant recipient.
* Patient is on any type of immunosuppression (i.e. prior transplant recipient still on immunosuppression, or patient is receiving systemic steroids for any medical condition).
* Patient, who, in the opinion of the investigator, has significant medical or psychosocial problems or unstable disease states which would preclude enrollment. Examples of significant medical problems include, but are not limited to, morbid obesity or severe cardiac disease.
* Kidneys that are to be implanted en bloc or from donors less than 6 years old.
* Kidneys from donors that are known or suspected to have an active infection with or be seropositive for HBsAg, hepatitis B core antibody (HBcAb), HCV, or HIV.
* Kidneys from donors that have received investigational therapies designed to reduce the impact of ischemia reperfusion, DGF, or other donor-related immune events.
* Donor kidney is preserved by cold storage (with or without machine preservation) for less than 16 hours, with the exception of kidneys from non-heart-beating donors or kidneys from donors greater than 50 years old or donors with a SCr above 2.5mg/dL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2000-05; Primary Completion 2003-04 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Freedom from acute rejection, kidney transplant loss, delayed kidney transplant function and death at 6 months after transplant. | 6 months

SECONDARY OUTCOMES:
12-mo. safety & efficacy assessments including side effects and overall kidney transplant function. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (28):
- United States (16):
  - University of Alabama, Birmingham, Alabama
  - UCLA School of Medicine, Los Angeles, California
  - California Pacific Medical Center, San Francisco, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Florida Hospital Medical Center and Translife, Orlando, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - Rush University Transplant Program, Chicago, Illinois
  - University of Kentucky Medical Center, Lexington, Kentucky
  - University of Michigan Hospital, Ann Arbor, Michigan
  - St. Barnabas Medical Center, Livingston, New Jersey
  - Westchester Medical Center, Valhalla, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Texas Medical Branch, Galveston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- France (5):
  - Hopital Saint Jacques, Besançon
  - Hopital de Bradois, Cedex
  - Centre Hospitalier Universitaire, Grenoble
  - Hopital Edouard Herriot, Lyon
  - Hopital Foch, Suresnes
- Germany (2):
  - Unicersitat Erlangen-Numberg, Erlangen
  - University Hospital Eppendorf, Hamburg
- Spain (4):
  - Hospital de Cruces, Barakaldo
  - Hospital Clinico Universitario, Barcelona
  - Hospital Reina Sofia, Córdoba
  - Hospital Occe de Octubre, Madrid
- Freeman Hospital, Newcastle upon Tyne, United Kingdom

REFERENCES:
- [Result] Brennan DC, Daller JA, Lake KD, Cibrik D, Del Castillo D; Thymoglobulin Induction Study Group. Rabbit antithymocyte globulin versus basiliximab in renal transplantation. N Engl J Med. 2006 Nov 9;355(19):1967-77. doi: 10.1056/NEJMoa060068. PMID 17093248
- [Derived] Lentine KL, Schnitzler MA, Xiao H, Brennan DC. Long-term safety and efficacy of antithymocyte globulin induction: use of integrated national registry data to achieve ten-year follow-up of 10-10 Study participants. Trials. 2015 Aug 19;16:365. doi: 10.1186/s13063-015-0891-y. PMID 26285695
- See also: US FDA Approved Full Prescribing Information for Thymoglobulin® — http://www.thymoglobulin.com/home/thymo_pdf_pi.pdf